CLINICAL TRIAL: NCT06019104
Title: Investigation of the Effects of Task-Oriented Training on Balance and Gait in Patients With Peripheral Vestibular Hypofunction
Brief Title: Effects of Task-oriented Training in Patients With Peripheral Vestibular Hypofunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Yasemin Apaydın, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25901600-604.01.01-12
Record Dates: First submitted 2021-12-07; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Peripheral Vestibular Disorders
Keywords: Task-oriented training; Balance; Gait; Vertigo; Dizziness; Quality of life
MeSH Terms: conditions — Vertigo; Dizziness | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task-oriented training group (Experimental): Among the patients in the task-oriented training group, 12 sessions were given routinely, 3 days a week, for 4 weeks. Task-oriented training consisted of 25 different stations in total, including 9 different gaze stabilization training, 7 balance training, and 9 gait training stations. Gaze stabilization exercises included head-fixed right-left eye movements, head-fixed up-down eye movements, eye fixed right-left head movements, eye fixed up-down head movements, head and eye opposing movements (right-left/ up-down), saccadic and pursuit eye movements (right-left/ up-down). Balance and gait training included these exercises: rolling on the mat, vertical rotation, spinning on a rotary disc, standing on balance bord, jumping, playing dart, reaching, walking forward, walking with head movements (right-left/ up-down), tandem walking, '8' shape walking, walking by picking something up from the ground, walking over an obstacle, walking on treadmill, climbing and descending stairs.
  Interventions: Other: Task-oriented training
- Control group (Active Comparator): Among the patients in the control group with peripheral vestibular disorders, 12 sessions were given routinely, 3 days a week, for 4 weeks. They were asked to perform gaze stabilization exercises for 1 min. Gaze stabilization exercises consist of head-fixed right-left eye movements, head-fixed up-down eye movements, eye fixed right-left head movements, and eye fixed up-down head movements.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Task-oriented training — Task-oriented training is defined as an approach based on movement science and motor learning, where the patient "makes functional movements specific to a certain task and receives feedback". Task-oriented training focuses on improving performance on functional tasks through targeted practice and repetition.
  Arms: Task-oriented training group
Other: Control group — Gaze stabilization exercises included head-fixed right-left eye movements, head-fixed up-down eye movements, eye fixed right-left head movements, and eye fixed up-down head movements.
  Arms: Control group

SUMMARY:
The peripheral vestibular disorder is a heterogeneous disorder that occurs due to unilateral or bilateral involvement of the peripheral vestibular organs in the inner ear, characterized by dizziness, balance disorder, visual blurring with head movements, postural instability, and gait disturbance. In the treatment of vestibular disorders, medical and surgical approaches, as well as vestibular rehabilitation are included. Vestibular rehabilitation should aim at repetitive stimulation of the vestibular sensory organs and improving peripheral sensory inputs by providing strong synaptic plasticity between the hair cells in these organs and the damaged parts of the vestibular system. According to this information, task-oriented training based on the practice of the task in the real environment with plenty of repetition seems to be a suitable method for the requirements of the treatment of vestibular disorders. This study was planned to examine the effects of task-oriented training on balance and gait in patients with peripheral vestibular disorders.

DETAILED DESCRIPTION:
Patients with peripheral vestibular disorders refrain from moving because of the increase in dizziness and fear of falling. These patients prefer to stay still and limit themselves even in simple daily life activities such as vacuuming, cleaning the table, and walking. From this point of view, it is thought that using the tasks in daily life or the activities that form the basis of these tasks in treatment as in task-oriented training will reduce the activity limitations caused by vestibular disorders.

In the recovery of the vestibular system, it is important to practice the functions that increase the symptoms with many repetitions. For example, symptoms that occur without head movement in the acute period after vestibular injury resolve rapidly, and disappear to a large extent as vestibular compensation develops. However, as the disease becomes chronic, losses occur in afferent inputs from the vestibular system and cause a negative effect on dynamic reflex functions. Therefore, vestibular rehabilitation should be aimed to stimulate the vestibular sensory organs repeatedly and to improve peripheral sensory inputs by providing strong synaptic plasticity between the hair cells in these organs and the damaged parts of the vestibular system. According to this information, task-oriented training based on the practice of the task in the real environment with plenty of repetition seems to be a suitable method for the requirements of the treatment of vestibular disorders.

In addition, there is evidence that task-oriented training improves balance, mobility, and gait reduces the risk of falls, and improves the quality of life in neurological diseases such as Stroke, Multiple Sclerosis, and Parkinson's disease. This information supports the investigators' idea that task-oriented training may also be beneficial in improving balance and walking performance, which are the main symptoms of peripheral vestibular disorder.

On the other hand, when the investigators examine the literature, there is no study examining the effects of task-oriented education in patients with peripheral vestibular disorders.

The primary aim of this study is to examine the effects of task-oriented training on vertigo, dizziness, balance, gait and falls in patients with peripheral vestibular disorders. The secondary aim of the investigators' study is to examine the effects of task-oriented training on disability level and quality of life in patients with peripheral vestibular disorders.

ELIGIBILITY:
Inclusion Criteria:

* Receiving a diagnosis of peripheral vestibular disorder by a specialist physician
* Being between the ages of 18-65
* Not having an inability to prevent the exercise
* Not having an Orthopedic, Neurological, Rheumatological, etc., which may cause balance disorder.

Exclusion Criteria:

* Having cognitive dysfunction that may affect the research results.
* Having a history of cerebrovascular accident, fainting, or epilepsy
* Being included in the vestibular rehabilitation program in the last 1 month
* Being in the acute phase of vestibular disease
* Having benign paroxysmal positional vertigo
* Using vestibular suppressant and centrally acting drugs in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Posturography | 4 weeks
  The posturography evaluation was made using the Synapsis Posturography System® (SPS®, version 3.0). All patients performed the Sensory Organization Test (SOT), this test representing the association between static and sway-referenced support in posturography under three conditions - eyes open (eo), eyes closed (ec), mislead vision. SOT objectively analyses the three sensory systems that contribute to postural control: somatosensory, visual and vestibular, by systematically eliminating useful visual or support information, creating also sensory conflict situations. We registered the results obtained under six conditions: eyes open, eyes closed and looking sway-referenced screen on static surface and sway-referenced surface. The feet position of the patient on the platform was - 2 cm spacing apart of the heels and a 30º angle between, corresponding to the foot size. Each test was performed barefoot, in standing position, 2 trials of 20 seconds for each test.
G-walk® spatio-temporal gait analysis system (speed) | 4 weeks
  The gait speed was assessed by G-walk® spatio-temporal gait analysis system. The assessment began with the participant standing still in an orthostatic standing position. The position had to be maintained for a few seconds until the end of the stabilization of the G-Walk device. The participants were instructed to walk on a 8 meter track. The boundaries of the track were marked to ensure a correct analysis. The participants walked at their natural speed along an absolutely straight path. A successful trial was characterized by the participant completing the 8-meter track and returning to the starting point. The parameter that were evaluated using the G-Walk were; speed (meter/seconds).This parameter are recorded by G-walk and transferred to the computer.
G-walk® spatio-temporal gait analysis system (cadence) | 4 weeks
  The cadence was assessed by G-walk® spatio-temporal gait analysis system. The gait assessments began with the standing position. The position had to be maintained for a few seconds until the end of the stabilization of the G-Walk device. On an 8 meter track, the participants were asked to walk. For a proper examination, the track's limits were delineated. The participants followed a perfectly straight line while moving at their usual pace. The participant's completion of the 8-meter track and arrival back at the starting point defined a successful trial. Cadence was the parameter that was assessed using the G-Walk.This parameter is sent to the computer after being recorded by G-walk.

SECONDARY OUTCOMES:
The severity and frequency of vertigo and dizziness (Visual analog scale (VAS)) | 4 weeks
  In order to evaluate the severity of vertigo and dizziness, the patients were shown a 12.5×17.5 cm Visual analog scale (VAS) card in which the expressions were written in 36 points. VAS was used to determine the severity of vertigo and dizziness. Patients were asked to rate 1=no vertigo/dizziness, 2-3=mild, 4-5=moderate, 6-7=severe, 8-9=very severe, and 10=extreme.
  In order to evaluate the frequency of vertigo and dizziness in the last 7 days, a 13×18 cm VAS scale card in which the expressions were written in 36 points was used. Patients were asked to rate; 1= no vertigo/dizziness, 2-3= 1-5 times a week, 4-5= 1-3 times a day, 6-7= 4-10 times a day, 8-9= >10 times a day, 10= continuous vertigo.
Disability level and quality of life | 4 weeks
  The Dizziness Handicap Inventory (DHI) evaluates the disability level and quality of life in patients with dizziness. The scale measures the functional, physical and emotional effects of dizziness in the last 1 month. The scale, which consists of 25 questions in total, has 3 subsections: physical (7 questions), emotional (9 questions) and functional (9 questions).
  The scale, which has 3 answer options as 'yes', 'sometimes' and 'no' for each question, has a score of 4, 2 and 0 for each answer, respectively. The maximum score is 100, with 28 for the physical subsection and 36 for the emotional and functional subsections. According to this; 0-30 points are indicated as light handicap; 30-60 points are indicated as moderate disability and 60-100 points are indicated as severe disability.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Güçlü-Gündüz, Prof, Study Director — Professor Doctor
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soke F, Guclu-Gunduz A, Kocer B, Fidan I, Keskinoglu P. Task-oriented circuit training combined with aerobic training improves motor performance and balance in people with Parkinson's Disease. Acta Neurol Belg. 2021 Apr;121(2):535-543. doi: 10.1007/s13760-019-01247-8. Epub 2019 Nov 18. PMID 31741209
- [Background] Ozkul C, Guclu-Gunduz A, Eldemir K, Apaydin Y, Gulsen C, Yazici G, Soke F, Irkec C. Effect of task-oriented circuit training on motor and cognitive performance in patients with multiple sclerosis: A single-blinded randomized controlled trial. NeuroRehabilitation. 2020;46(3):343-353. doi: 10.3233/NRE-203029. PMID 32310197
- [Background] Tramonti C, Di Martino S, Chisari C. An intensive task-oriented circuit training positively impacts gait biomechanics in MS patients. NeuroRehabilitation. 2020;46(3):321-331. doi: 10.3233/NRE-192997. PMID 32250333
- [Background] Kim B, Park Y, Seo Y, Park S, Cho H, Moon H, Lee H, Kim M, Yu J. Effects of individualized versus group task-oriented circuit training on balance ability and gait endurance in chronic stroke inpatients. J Phys Ther Sci. 2016 Jun;28(6):1872-5. doi: 10.1589/jpts.28.1872. Epub 2016 Jun 28. PMID 27390437
- [Background] Arnold SA, Stewart AM, Moor HM, Karl RC, Reneker JC. The Effectiveness of Vestibular Rehabilitation Interventions in Treating Unilateral Peripheral Vestibular Disorders: A Systematic Review. Physiother Res Int. 2017 Jul;22(3). doi: 10.1002/pri.1635. Epub 2015 Jun 25. PMID 26111348
- [Background] Hillier S, McDonnell M. Is vestibular rehabilitation effective in improving dizziness and function after unilateral peripheral vestibular hypofunction? An abridged version of a Cochrane Review. Eur J Phys Rehabil Med. 2016 Aug;52(4):541-56. Epub 2016 Jul 12. PMID 27406654